CLINICAL TRIAL: NCT00619593
Title: Survival of Patients With Primary Prophylactic ICD Indication, Provided With Intensified Care After 1st ICD Therapy
Brief Title: Survival of Patients With Primary Prophylactic ICD Indication
Acronym: SPIRIT-ICD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TA079
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Primary Prevention; Tachycardia, Ventricular; Sudden Cardiac Death
Keywords: Heart failure; Ventricular Fibrillation; Sudden cardiac death; Hospitalization due to heart failure; Implantable cardioverter-defibrillator; Risk of 1st heart failure hospitalization
MeSH Terms: conditions — Tachycardia, Ventricular; Death, Sudden, Cardiac; Heart Failure; Ventricular Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): Standard follow-up in patients without appropriate ICD therapy
  Interventions: Other: Standard follow-up
- 1 (Experimental): Following 1st appropriate ICD therapy, the patients have to be called to the clinic for intensified clinical diagnostics and, if necessary or useful, intensified therapy.
  Interventions: Other: Intensified diagnostic and treatment measures following 1st appropriate ICD therapy

INTERVENTIONS:
Other: Intensified diagnostic and treatment measures following 1st appropriate ICD therapy — * Assessment of general health status (weight, BP, NYHA)
  * Laboratory tests (hemoglobin, Nt-proBNP, creatinine, GDF-15)
  * Echocardiography (LVEF, LVEDD, mitral regurgitation)
  * Non-invasive ischemia evaluation
  * Coronary angiography (if indicated by ischemia evaluation)
  * Upgrade to CRT, if indicated
  * Ventricular ablation (if indicated: VT storm, slow VT, bundle branch reentry)
  * 24 hrs ECG Holter (Heart rate variability)
  * Further treatment (if applicable)
  * Changes in ICD settings, or medication
  Other Names: Intensified diagnostic and treatment measures
  Arms: 1
Other: Standard follow-up — Standard follow-up in patients without appropriate ICD therapy
  Arms: 2

SUMMARY:
The MADIT-II trial has shown that patients with severely reduced left ventricular ejection fraction (LVEF) post myocardial infarction benefit from the implantable cardioverter-defibrillator (ICD). However, retrospective analyses of the MADIT-II data have revealed a significantly increased morbidity and mortality in patients with appropriate ICD therapy: Appropriate ICD therapy is associated with 3.3-fold increased all-cause mortality, and the risk of a first heart failure hospitalization is 90% higher after 1st appropriate ICD therapy. Hence, the 1st appropriate therapy might indicate the necessity and utility of further clinical diagnostics and therapy in these patients.

This trial is designed to (i) improve the knowledge of the group characteristics of patients suffering from 1st appropriate ICD therapy, (ii) but moreover to take additional therapeutic steps to reduce the mortality of this patient population.

DETAILED DESCRIPTION:
The MADIT-II trial has shown that patients with severely reduced left ventricular ejection fraction (LVEF) post myocardial infarction benefit from the implantable cardioverter-defibrillator (ICD). However, retrospective analyses of the MADIT-II data have revealed a significantly increased morbidity and mortality in patients with appropriate ICD therapy: Appropriate ICD therapy is associated with 3.3-fold increased all-cause mortality, and the risk of a first heart failure hospitalization is 90% higher after 1st appropriate ICD therapy. Hence, the 1st appropriate therapy might indicate the necessity and utility of further clinical diagnostics and therapy in these patients.

This trial is designed to (i) improve the knowledge of the group characteristics of patients suffering from 1st appropriate ICD therapy, (ii) but moreover to take additional therapeutic steps to reduce the mortality of this patient population.

After standard ICD implantation procedure, the following steps are performed at the pre-discharge follow-up:

* Programming: VR-T: VVI 40 ppm, Onset 20%, Stability 20 ms
* DR-T: DDD 50-60 ppm, activation of IRSplus and SMART
* HF-T: DDD-BiV 50-60 ppm, achieve at least 85% biventricular resynchronisation, activation of SMART
* All devices: VT zone as therapy zone, VF zone. Programming recommendations for VT/VF zones to standardize treatment:

  * VF zone: 200-250 bpm/ 300-240 ms, ATPoneshot ON
  * VT1 zone: 167-200 bpm/ 360-300 ms, ATP ON
  * VT2 zone: 120-167 bpm/ 500-360 ms, ATP ON
* Activation of Home Monitoring (HM) and online registration for HM service

Standard Follow-up: Timing and scope of follow-up in patients without episodes is to the physician's own discretion and should follow the standard clinical routine.

Follow-up after 1st appropriate ICD therapy: Immediately after having received the 1st appropriate ICD therapy, the patients have to be called to the clinic for intensified clinical diagnostics and, if necessary or useful, intensified therapy. Standard ICD follow-up has to be started within 72 hours after 1st appropriate ICD therapy.

* ICD interrogation
* General health status (weight, BP, NYHA)
* Laboratory tests (hemoglobin, Nt-proBNP, creatinine, GDF-15)
* Echocardiography (LVEF, LVEDD, mitral regurgitation)
* Non-invasive ischemia evaluation
* Coronary angiography (if indicated by ischemia evaluation)
* Upgrade to CRT, if indicated
* Ventricular ablation (if indicated: VT storm, slow VT, bundle branch reentry)
* 24 hrs ECG Holter (Heart rate variability)
* Further treatment (if applicable)
* Changes in ICD settings, or medication
* Adverse events / adverse device effects

Final follow-up visit: For patients without appropriate ICD therapy, the final follow-up shall be performed 12 months after enrolment.

For patients with appropriate ICD therapy, the final follow-up shall be performed 12 months after 1st appropriate ICD therapy.

The final follow-up visit comprises:

* ICD interrogation
* General health status (weight, BP, NYHA)
* Echocardiography (LVEF, LVEDD, mitral regurgitation)
* Laboratory tests (hemoglobin, Nt-proBNP, creatinine, GDF-15)
* 24 hrs ECG Holter (Heart rate variability)
* Further treatment (if applicable)
* Changes in ICD settings, or medication
* Adverse events / adverse device effects

ELIGIBILITY:
Inclusion Criteria:

* Indication for ICD implantation according to MADIT-II:

  * Myocardial infarction 30 days or more before implantation
  * LVEF of 30% or less within 3 months before implantation
* Angiography within the preceding 12 months
* The patient is willing and able to comply with the clinical investigation plan and has provided written informed consent

Exclusion Criteria:

* Patients with contraindication for ICD implantation
* Conventional ICD indication (i.e. other than MADIT-II)
* Myocardial infarction within the past 30 days
* Coronary revascularisation within the preceding 3 months (i.e., if revascularization has been performed wait at least 3 months until enrolment, given that no appropriate/ inappropriate ICD therapy has occured)
* NYHA functional class IV
* Unexplained syncope within 3 years
* Advanced cerebrovascular disease
* Life expectancy very probably below 12 months
* Pregnant or breast-feeding women
* Age < 18 years
* Patients who are already enrolled in another study (therapy/intervention phase)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2008-02; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Mortality | 12 months

SECONDARY OUTCOMES:
Sudden cardiac death | 12 months
Non-sudden cardiac death | 12 months
Risk of 1st heart failure hospitalization | 12 months
No. of VT Storms (> 3 VT/24h) | 12 months
No. of delivered ICD therapies | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hatala, Prof. MUDr., Principal Investigator — Národný ústav srdcových a cievnych chorôb, Kardiologická klinika, Pod Krásnou Hôrkou 1, 833 48 Bratislava, Slovakia
Locations (37):
- Austria (3):
  - A.ö. Krankenhaus der Stadt Linz, Linz
  - Landesklinikum St. Pölten, Sankt Pölten
  - Wilhelminenspital der Stadt Wien, Vienna
- Czechia (5):
  - Brno Bohunice, Brno
  - Fakultni nemocnice u Svety Anny, Brno
  - FN Olomouc, Inerni klinika, Olomouc
  - Online 24 S.R.O., Prague
  - Institute of clinical and experimental medicine, Prague
- Germany (17):
  - University Hospital RWTH Aachen, Aachen
  - Herz- und Gefäss-Klinik GmbH Bad Neustadt, Bad Neustadt an der Saale
  - Klinikum Bielefeld, Bielefeld
  - Universitätsklinikum Bonn, Bonn
  - St. Marien Hospital, Bonn
  - Klinikum Detmold Lippe, Detmold
  - Klinikum Mitte, Dortmund
  - Städtisches Klinikum Dresden-Friedrichstadt, Dresden
  - Evangelisches Krankenhaus, Düsseldorf
  - Hermann-Josef-Krankenhaus, Erkelenz
  - Justus Liebig Universität Gießen, Giessen
  - Medizinische Hochschule Hannover, Hanover
  - Krankenhaus Landshut-Achdorf, Landshut
  - Krankenhaus St. Franziskus, Mönchengladbach
  - St. Vincenz Krankenhaus, Paderborn
  - University Hospital Rostock, Rostock
  - Katharinenhospital, Unna
- Hungary (2):
  - Semmelweis University, Budapest
  - The University of Medicine Debrecen, Debrecen
- Chaim Sheba Medical Center, Tel Litwinsky, Israel
- Latvian Center of Cardiology, Riga, Latvia
- Health Waikato, Cardiology Department, Hamilton, New Zealand
- Poland (2):
  - MULTI-MED PLUS Spolka z o.o, Lodz
  - Instytut Kardiologii, Warzawa
- Slovakia (3):
  - Ssusch, Banská Bystrica
  - Kardiologická klinika, Bratislava
  - VUSCH East Slovak Cardiology Institute, Košice
- H. Univ. La Fe, Valencia, Spain
- Universitätsspital Basel, Basel, Switzerland